CLINICAL TRIAL: NCT06055868
Title: People Living With HIV (PLWH), Oral and Oropharyngeal Cancer, and Health Equity: A Qualitative Study
Brief Title: People Living With HIV, Oral and Oropharyngeal Cancer, and Health Equity
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23363; R03DE032972 (NIH)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections; Oral Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
Keywords: Health Equity; Focus Group; Sexual and Gender Minority; People living with HIV; HPV, human papillomavirus
MeSH Terms: conditions — HIV Infections; Squamous Cell Carcinoma of Head and Neck; Coitus; Papillomavirus Infections | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative Focus Group: Participants will be asked to a series of questions to help place them in a focus group with other individuals of shared identity and will also complete a short quantitative survey either emailed to the participant or the outreach worker/study coordinator will administer the survey by phone. Participants will then participate in one 1.5-2 hour, facilitated, focus group discussions (FGD).
  Interventions: Other: Group Meeting (Focus Group); Other: Questionnaires

INTERVENTIONS:
Other: Group Meeting (Focus Group) — Focus Group Discussions (FDGs) will be recorded, transcribed, and coded.
Other: Questionnaires — Given electronically or via phone by study team staff

SUMMARY:
This is an exploratory qualitative study among People Living With HIV (PLWH) of diverse racial/ethnic and sexual and gender minority (SGM) identities to explore individual, interpersonal, and structural oral health equity factors that serve as barriers or facilitators of accessing oral health care, knowledge and perceptions of human papillomavirus (HPV) vaccination and Oral squamous cell carcinoma (OSCC) /Oropharyngeal squamous cell carcinoma (OPSCC), and to collect recommendations on how to increase access to oral health care and engage PLWH in OSCC/OPSCC prevention.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To identify individual, interpersonal, and structural oral health equity factors (e.g., internalized stigma; enacted stigma; transportation/hours) that serve as barriers or facilitators to accessing regular and appropriate oral health care, among PLWH of intersecting racial/ethnic and SGM groups.
2. To explore knowledge and perceptions about causes, risk factors, prevention, and screening for OSCC/OPSCC and HPV vaccination and if identity group membership influences knowledge and perceptions of these issues.
3. To elicit recommendations for improving access to regular and appropriate oral health care, and suggestions on how to engage PLWH from diverse identity groups in prevention interventions.

OUTLINE:

There will be one screening and enrollment phone call and only one study visit for the Focus Group Discussions (FDGs). A short quantitative survey will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-years old or older.
* Participants must be individuals living with HIV
* Ability to speak and understand English
* Identify as one or more racial/ethnic minority groups or sexual and gender minority groups
* All genders and members of all races and ethnic groups are eligible for this study.

Exclusion Criteria:

* Younger than 18-years old.
* Not living with HIV.
* Not able to speak and understand English.
* Not classified as one or more racial/ethnic minority groups or sexual and gender minority groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV who identify with one or more racial/ethnic/ sexual or gender minority groups
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of potential oral health equity factors | Up to 3 days
  Participants will complete a baseline questionnaire which will aid in the formation of the focus group with other individuals of shared identity. The Focus Group Discussions (FGDs) will be transcribed, coded, and the focus group guide will be updated following the Grounded Theory qualitative research methodology. The "data" from the FGD are the audio recordings and the transcripts. The digital transcript of each focus group will be uploaded to the software MAXQDA to aid with coding and analysis in identifying individual, interpersonal, and structural factors, if any, that may impact accessing oral health care.

OTHER OUTCOMES:
Assess participant perceptions about OSCC/OPSCC and HPV vaccination | During focus group, 1 day
  FGDs will be transcribed, coded, and the focus group guide will be updated following the Grounded Theory qualitative research methodology. The "data" from the FGD are the audio recordings and the transcripts. The digital transcript of each focus group will be uploaded to the software MAXQDA to aid with coding and analysis in assessing information on participant's perception of causes, risk factors, prevention, and screening for OSCC/OPSCC and HPV vaccination.
Assess participant knowledge about OSCC/OPSCC and HPV vaccination | During focus group, 1 day
  FGDs will be transcribed, coded, and the focus group guide will be updated following the Grounded Theory qualitative research methodology. The "data" from the FGD are the audio recordings and the transcripts. The digital transcript of each focus group will be uploaded to the software MAXQDA to aid with coding and analysis in assessing information on participant's knowledge of causes, risk factors, prevention, and screening for OSCC/OPSCC and HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Hernandez Levenston, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez AL, Lingas EO, Juarez W, Villa A, Palefsky J. Using an anti-racist research framework to design studies of oral human papillomavirus and oropharyngeal cancer in San Francisco: rationale and protocol for the Health Equity and Oral Health in People living with HIV (HEOHP) qualitative study. BMJ Open. 2024 Sep 24;14(9):e091474. doi: 10.1136/bmjopen-2024-091474. PMID 39317508